CLINICAL TRIAL: NCT01052493
Title: A First Time in Human, Double Blind, Randomised, Placebo Controlled Dose Escalation Study to Assess the Safety and Tolerability of PP 1420 in Healthy Subjects.
Brief Title: A First-Time-in-Human Study to Assess the Safety and Tolerability of PP 1420 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Wellcome Trust (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ICIM1420/09/01; 2009-017522-39 (EudraCT Number)
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Results first posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: obesity; pancreatic polypeptide; gut hormones
MeSH Terms: conditions — Obesity | interventions — PP 1420; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: There were three dosing periods. Each subject (n=12) was randomised to receive up to two doses of placebo and/or up to three ascending doses of PP 1420 dosed as s.c. injection. During each dosing period eight subjects received active drug and four received placebo. Subjects could also be randomised to receive one further dose of PP 1420 or placebo, if needed, to explore an intermediate dose based upon a review of safety, tolerability, and PK data from the previous cohorts.
Who Masked: Participant, Investigator
Masking Description: This was a double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2mg PP 1420 (Experimental): PP 1420 single dose, subcutaneous
  Interventions: Drug: PP 1420
- 4mg PP 420 (Experimental): PP 1420 single dose, subcutaneous
  Interventions: Drug: PP 1420
- 8mg PP 1420 (Experimental): PP 1420 single dose, subcutaneous
  Interventions: Drug: PP 1420
- Placebo (Placebo Comparator): 0.9% saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PP 1420 — Single dose of PP 1420, administered subcutaneously at either 2mg, 4mg or 8mg.
  Other Names: PP 1420 pancreatic polypeptide analog
  Arms: 2mg PP 1420; 4mg PP 420; 8mg PP 1420
Drug: Placebo — 0.9% saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
When humans eat, the bowels naturally secrete chemicals into the bloodstream which make people feel full and which stop eating. One of these chemicals is known as "Pancreatic Polypeptide" (PP). We have previously shown that injections of human PP reduces appetite and food intake. We have now developed a very similar chemical, PP 1420, as a treatment for obesity. PP 1420 has been tested in animals and has been shown to be safe, and to reduce their appetite. This study will test PP 1420 for its safety and tolerability in humans.

DETAILED DESCRIPTION:
More than 20 percent of people in the UK are obese. People with obesity have a shorter life expectancy, and have a higher risk of having heart attacks, strokes, high blood pressure, diabetes, and certain cancers.

At the moment, there is no treatment for obesity that is both effective and safe. Advising people to change their diet and to exercise more is frequently ineffective, and any loss in weight seen is usually temporary. There are a couple of licensed medications for the purpose of losing weight, but they are limited by side effects. Finally, gastric bypass and similar surgeries are effective at reducing weight permanently, but it can be risky and is restricted only to very motivated people.

"Gut hormones" are natural chemicals made by the bowels when you eat. They work to reduce appetite and hunger when you eat, so that you will eat enough for your needs. We think that one of the reasons why gastric bypass surgery is so effective is because the surgery causes an increase in gut hormone secretion into the bloodstream, which suppresses appetite. One of these hormones is pancreatic polypeptide (PP), which is released into the bloodstream by cells in the pancreas after eating. When human PP is given to healthy volunteers as an injection, we see that they have a reduced appetite and food intake with no side effects such as feeling sick or vomiting.

Human PP does not last long in the blood stream. In order to make it into a new, safe and effective drug for obesity, we have developed a new form of PP, which is very similar but not identical to human PP, that we expect will last longer in the blood. We call this PP 1420.

In testing, PP 1420 reduced food intake in animals, and was safe in them at much higher doses than those we plan to give in the current study. This study will assess the safety and tolerability of PP 1420 in humans, and is the first time humans have been given this medication.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male as determined by a responsible physician, based on a medical evaluation including history, physical examination, vital signs, laboratory tests and 12-lead ECG.
* Between 18 and 50 years of age, inclusive, at the time of signing and dating the informed consent form.
* Body weight ≥70 kg and body mass index (BMI) within the range 18 - 35 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Willing and able to comply with the protocol for the duration of the study.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unsuitable for the study.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for human immunodeficiency virus (HIV) antibody.
* History of migraine.
* History or evidence of abnormal eating behaviour, as observed through the Dutch Eating Behaviour (DEBQ) and SCOFF questionnaires.
* History of excessive alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units. One unit is equivalent to 8 g of alcohol, a half-pint (approximately 240 mL) of beer or 1 measure (25 mL) of spirits or 1 glass (125 mL) of wine.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Has QTc at screening >450 msec.
* Systolic blood pressure outside the range 85 - 160 mmHg, diastolic blood pressure outside the range 45 - 100 mmHg, and/or heart rate outside the range 40 - 110 bpm.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the dosing day in the current study: 90 days, five half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or five half-lives (whichever is longer) prior to the dose of study medication, which, in the opinion of the Investigator, may interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator, contraindicates their participation.
* Where participation in the study would result in donation of blood in excess of 500 mL within 3 months before or after the study.
* Unwilling to abstain from consumption of caffeine- or xanthine- containing products for 24 hours prior to dosing until the post-dose assessment at each treatment level.
* Unwilling to abstain from use of illicit drugs.
* Unwilling to abstain from alcohol for 48 hours prior to dosing until final post-dose assessment at each treatment level.
* Unwilling to abstain from smoking or otherwise consuming tobacco for 24 hours prior to dosing until the post-dose assessment at each treatment level.
* Unwilling to use a condom during sexual activity from first dose until the end of the study.
* Vegans and subjects with milk or wheat intolerance or allergy as reported by the subject.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male
Enrollment: 13 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2010-10-18 (Actual); Study Completion 2010-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bloom FRCP DSc, MB BChir, Principal Investigator — Imperial College London
Locations (1):
- Sir John McMichael Centre for Clinical Studies, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batterham RL, Le Roux CW, Cohen MA, Park AJ, Ellis SM, Patterson M, Frost GS, Ghatei MA, Bloom SR. Pancreatic polypeptide reduces appetite and food intake in humans. J Clin Endocrinol Metab. 2003 Aug;88(8):3989-92. doi: 10.1210/jc.2003-030630. PMID 12915697
- [Background] Jesudason DR, Monteiro MP, McGowan BM, Neary NM, Park AJ, Philippou E, Small CJ, Frost GS, Ghatei MA, Bloom SR. Low-dose pancreatic polypeptide inhibits food intake in man. Br J Nutr. 2007 Mar;97(3):426-9. doi: 10.1017/S0007114507336799. PMID 17313701
- [Result] Tan TM, Field BC, Minnion JS, Cuenco-Shillito J, Chambers ES, Zac-Varghese S, Brindley CJ, Mt-Isa S, Fiorentino F, Ashby D, Ward I, Ghatei MA, Bloom SR. Pharmacokinetics, adverse effects and tolerability of a novel analogue of human pancreatic polypeptide, PP 1420. Br J Clin Pharmacol. 2012 Feb;73(2):232-9. doi: 10.1111/j.1365-2125.2011.04082.x. PMID 21834938

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at Sir John McMichael Centre, Hammersmith Hospital
Pre-assignment Details: 12 participants started the study. It was a sequential cross-over study. They were randomised to receive either PP 1420 or placebo at each treatment stage. After the first treatment period, one volunteer withdrew. This participant was replaced with a new participant in order that 12 participants progressed onto intervention periods 2 and then 3.
Groups:
- Placebo, 4mg PP 1420, 8mg PP 1420: Intervention Period 1: Placebo Intervention period 2: 4mg PP 1420 Intervention period 3: 8mg PP 1420
- 2mg PP 1420, Placebo, 8mg PP 1420: Intervention Period 1: 2mg PP 1420 Intervention Period 2. Placebo Intervention Period 3. 8mg PP 1420
- 2mg PP 1420, 4mg PP 1420, Placebo: Intervention Period 1: 2mg PP 1420 Intervention Period 2. 4mg PP 1420 Intervention Period 3. Placebo
Period: Intervention 1 (Up to 10 Days)
Arm/Group | Placebo, 4mg PP 1420, 8mg PP 1420 | 2mg PP 1420, Placebo, 8mg PP 1420 | 2mg PP 1420, 4mg PP 1420, Placebo
Started | 4 | 4 | 4
Completed | 3 | 4 | 4
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Washout Period 1 (up to 5 Days)
Arm/Group | Placebo, 4mg PP 1420, 8mg PP 1420 | 2mg PP 1420, Placebo, 8mg PP 1420 | 2mg PP 1420, 4mg PP 1420, Placebo
Started | 3 | 4 | 4
Completed | 3 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Intervention 2 (up to 10 Days)
Arm/Group | Placebo, 4mg PP 1420, 8mg PP 1420 | 2mg PP 1420, Placebo, 8mg PP 1420 | 2mg PP 1420, 4mg PP 1420, Placebo
Started | 4 (Replacement subject recruited) | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Washout Period 2 (up to 5 Days)
Arm/Group | Placebo, 4mg PP 1420, 8mg PP 1420 | 2mg PP 1420, Placebo, 8mg PP 1420 | 2mg PP 1420, 4mg PP 1420, Placebo
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Intervention 3 (up to 10 Days)
Arm/Group | Placebo, 4mg PP 1420, 8mg PP 1420 | 2mg PP 1420, Placebo, 8mg PP 1420 | 2mg PP 1420, 4mg PP 1420, Placebo
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The population of participants which started in dosing period 1
Groups:
- All Participant: Crossover, sequential study with all participant
Arm/Group | All Participant
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs)
Description: Number of subjects with adverse events recorded through the trial period
Time Frame: 7-12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- 2mg PP 1420; 4mg PP 1420; 8mg PP 1420: Single dose of PP 1420, administered subcutaneously
Arm/Group | 2mg PP 1420 | 4mg PP 1420 | 8mg PP 1420 | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 12
Participants
  Total number of AEs | 2 | 5 | 3 | 2
  Serious TEAEs | 0 | 0 | 0 | 0
  TEAEs leading to discontinuation | 0 | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0

2. Secondary Outcome: AUC0-t(Last)
Description: The area under the concentration vs. time curve of PP 1420 from time zero to the last sampling time, calculated by the linear trapezoidal rule
Time Frame: 24 hours
Population: PP 1420 arms only
Measure: Geometric Mean (Full Range); unit: ng ml-1 h
Arm/Group | 2mg PP 1420 | 4mg PP 1420 | 8mg PP 1420
Number analyzed (Participants) | 8 | 8 | 8
ng ml-1 h | 93.6 [49.7 to 126] | 229 [107 to 316] | 403 [205 to 589]

3. Secondary Outcome: AUC0-∞
Description: the area under the concentration vs. time curve for PP 1420, estimated from time zero to infinity
Time Frame: 24 hours
Population: PP 1420 arms only
Measure: Geometric Mean (Full Range); unit: ng ml-1 h
Arm/Group | 2mg PP 1420 | 4mg PP 1420 | 8mg PP 1420
Number analyzed (Participants) | 8 | 8 | 8
ng ml-1 h | 101 [67.6 to 131] | 241 [109 to 356] | 418 [210 to 600]

4. Secondary Outcome: Maximum Observed Plasma Drug Concentration (Cmax)
Time Frame: Within 24 hours
Population: PP 1420 arms only
Measure: Geometric Mean (Full Range); unit: ng ml-1
Arm/Group | 2mg PP 1420 | 4mg PP 1420 | 8mg PP 1420
Number analyzed (Participants) | 8 | 8 | 8
ng ml-1 | 26.3 [15.9 to 39.1] | 55.1 [37.5 to 74.2] | 95.7 [74.2 to 126]

5. Secondary Outcome: Time of Maximum Observed Concentration (Tmax)
Time Frame: Within 24 hours
Population: PP 1420 arms only
Measure: Median (Full Range); unit: hours
Arm/Group | 2mg PP 1420 | 4mg PP 1420 | 8mg PP 1420
Number analyzed (Participants) | 8 | 8 | 8
hours | 0.875 [0.32 to 2.00] | 1.00 [0.75 to 1.50] | 1.00 [0.50 to 1.50]

6. Secondary Outcome: Terminal Elimination Half-life (t½)
Description: Calculated from log 2/λz where λz is the apparent terminal rate constant.
Time Frame: Within 24 hours
Population: PP 1420 arms only
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | 2mg PP 1420 | 4mg PP 1420 | 8mg PP 1420
Number analyzed (Participants) | 8 | 8 | 8
hours | 2.42 [1.64 to 3.38] | 2.49 [1.69 to 3.60] | 2.61 [2.13 to 3.95]

ADVERSE EVENTS:
Time Frame: 7-12 weeks
Arm/Group | 2mg PP 1420 | 4mg PP 1420 | 8mg PP 1420 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 2/8 | 5/8 | 3/8 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2mg PP 1420 (N=8) | 4mg PP 1420 (N=8) | 8mg PP 1420 (N=8) | Placebo (N=12)
Headache (Nervous system disorders) | 1 (2) | 2 (2) | 1 (1) | 2 (2)
Injection site reaction/bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain/bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected finger (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold sore (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No